CLINICAL TRIAL: NCT04633655
Title: International Chemotherapy Induced Peripheral Neurotoxicity (CIPN) Assessment and Validation Study
Brief Title: International CIPN Assessment and Validation Study
Acronym: ICAVS
Status: Recruiting | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: ICAVS
Record Dates: First submitted 2020-06-09; First posted 2020-11-18 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy; Quality of Life
Keywords: clinimetrics; biomarker; PRO; outcome measures
MeSH Terms: interventions — Outcome Assessment, Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples for neurofilament light chain detection
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who are receiving a neurotoxic chemotherapy: List of neurotoxic drugs eligible for enrolment
  * Platinum drugs
  * Taxanes
  * Vinca alkaloids
  * Epothilones
  * Proteasome inhibitors
  * Thalidomide
  * Vedotin-based drugs
  * checkpoint inhibitors
  * Any combination of the aforementioned drugs
  Interventions: Other: outcome measures for CIPN testing

INTERVENTIONS:
Other: outcome measures for CIPN testing — questionnaires administration, physician based scales for CIPN data collection

SUMMARY:
This is an observational study of chemotherapy-induced peripheral neurotoxicity (CIPN) patients to be investigated prospectively in order to assess responsiveness of a set of outcome measures in an international multi-center study.

DETAILED DESCRIPTION:
The study will be performed at all participating centers and will consist of the following assessments:

Core study (assessments at baseline and at the end of treatment)

* Standard oncology assessment per local site
* NCI-CTC (national cancer institute common toxicity criteria) v.5 sensory and motor
* PRO-CTCAE (patient reported outcome-cancer common tocixity adverse event)
* PI-NRS (pain intensity numeric rating scale)
* NPS-CIN (Neuropathic Pain Scale for chemotherapy-induced neuropathy)
* EORTC CIPN20© (The European Organisation of Research and Treatment of. Cancer Quality of Life Questionnaire-CIPN twenty-item scale)
* FACT-GOG NTX v.4© (Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity)
* TNSn© (total neuropathy score, nurse version)
* PGIC (patient global impression of change)
* OXA-NQ (oxaliplatin neurotoxicity questionnaire)

Extended study (at all available sites - any combination of assessment methods is allowed, minimum at baseline and at the end of treatment)

* EORTC CIPN15
* CIPN-R-ODS (CIPN Rash overall disability scale)
* TNSc© at the same time points as for questionnaire
* OXA-NQ (also at mid-treatment)
* nerve conduction study of the radial (motor and sensory), ulnar (motor and sensory), sural, dorsal sural and common peroneal nerves (*)
* QST (*) [quantitative sensory testing]
* Serum for biomarkers search (*)
* DN4

Rationale: Within a multi-center international collaboration among experienced neurologists, oncologists, nurses and symptom scientists, the principal aim of this study is to evaluate responsiveness of a set of outcome measures for CIPN evaluation in order to define the gold standard for its assessment.

The assessment of CIPN will be performed at different levels of investigation. The Core study will allow the evaluation of subjects with common devices, so that an assessment can be performed at any medical site (expected time for questionnaires completion 15 minutes).

The Extended study will add any combination of the listed assessment methods/biological sample collection, in order to ascertain whether this approach can provide a more careful and clinically-relevant estimate of the peripheral nervous system damage. Comparison between healthcare evaluation and subjects' report of CIPN severity using established questionnaires will be performed in both Core and Extended studies.

Aims: The primary aim for this study is to test responsiveness of the different assessment methods used in the core study, in a multi-center, multi-regional International setting, comparing changes from baseline to end of treatment. Secondary aims are:

* to evaluate responsiveness (changes from base line to end of treatment) also of the other outcome measures used in the Extended Study;
* to evaluate mid-treatment data predictiveness of end of treatment neurological status for each outcome measure;
* to evaluate recovery rate/modification of the neurological status for the follow up evaluations (3/6/12/24 months after treatment), stratifying data for different drugs.

Study Design: 1000 patients who are candidates for neurotoxic chemotherapy for any cancer with non-investigational drugs (including immune checkpoint inhibitors and "targeted" drugs) will be enrolled from participating centers. A trained investigator in each participating center will perform the selected healthcare-assessed scales and supervise the patient-completed measures as presented in Table 1. Subjects will be examined at least at baseline and end of treatment (Core Study) and at additional intermediate and follow-up timepoints (Extended study), according to their treatment plan.

Study Treatments: There are no study-specified treatments, as subjects will receive only their standard of care chemotherapy. The investigators will not influence decisions regarding treatment duration nor supply medication for this study. However, all treatment regimens will be registered.

Participating Centers minimum requirements: Participating Centers should:

1. accept the study protocol and have their participation approved by a local Ethics Committee/Institutional Review Board
2. have access through an internet connection to the secure server located at the main site
3. guarantee the proper assessment of the selected patients at least at the Core study level
4. have the potential to recruit at least 30 patients/year
5. have the capacity to upload the data collected from each patient within 1 week

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following inclusion criteria to be eligible for enrolment into the study:

1. Subjects must be candidates for neurotoxic chemotherapy at doses expected to be potentially neurotoxic (a list of neurotoxic drugs is provided in Appendix 1).
2. Male and female subjects who are 18 years of age or older.
3. Subjects freely provide informed consent by signing and dating an informed consent form prior to study entry.
4. Subjects must be willing to complete all study-related activities and follow-up visits required by the protocol.
5. Subjects must have a Karnofsky performance score greater than or equal to 70. Exclusion Criteria

Subjects presenting with any of the following will not be included in the study:

1. Poor prognosis, with high probability to be unable to complete the planned chemotherapy treatment.
2. Concomitant neurologic conditions (e.g., brain tumor, spinal or brain metastases) that would interfere or complicate the assessments.
3. Severe depression that in the opinion of the Investigator would complicate the assessments.
4. Chronic treatment with antiepileptic drugs, antidepressants and major analgesics, unless stable dosing and conditions have been reached for 3 months prior to entry.
5. Preventive interventions (e.g., antioxidants, cryotherapy, distal pressure).
6. Subjects who are currently receiving another medication other than antineoplastic chemotherapy drugs that has known potential to produce neurologic peripheral nerve toxicity (e.g. metronidazole, isoniazid, amiodarone, antiretroviral medications).
7. Subjects with any other condition, which, in the investigator's judgment, might decrease the chance of obtaining satisfactory data to achieve the objectives of the study.
8. Previous neurotoxic chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients candidated to neurotoxic chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-06-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Chemotherapy-induced peripheral neurotoxicity as assessed by change in NCI-CTC v.5 sensory and motor grade | 5 YEARS
  NCI-CTC v.5 sensory and motor (changes from base line to end treatment of a 0-5 score)
Chemotherapy-induced peripheral neurotoxicity as assessed by change in PRO-CTCAE | 5 YEARS
  PRO-CTCAE (changes from base line to end treatment of a 0-5 score for each item)
Chemotherapy-induced peripheral neurotoxicity as assessed by change in Pain Intensity Numerical Rating Scale (PI-NRS) | 5 YEARS
  difference between baseline and end of treatment of chemotherapy-induced peripheral neurotoxicity as assessed by change in Pain Intensity Numerical Rating Scale (PI-NRS) (0-10 score).
Chemotherapy-induced peripheral neurotoxicity as assessed by change in NPS-CIN scale | 5 YEARS
  difference between baseline and end of treatment of chemotherapy-induced peripheral neurotoxicity as assessed by change in NPS-CIN (changes from base line to end treatment of a 0-10 score)
Chemotherapy-induced peripheral neurotoxicity as assessed by change in EORTC CIPN20© scale | 5 YEARS
  difference between baseline and end of treatment of chemotherapy-induced peripheral neurotoxicity as assessed by change in EORTC CIPN20© (changes from base line to end treatment of a 0-100 score)
Chemotherapy-induced peripheral neurotoxicity as assessed by change in FACT-GOG NTX v.4© scale | 5 YEARS
  difference between baseline and end of treatment of chemotherapy-induced peripheral neurotoxicity as assessed by change in FACT-GOG NTX v.4© (changes from base line to end treatment of a 0-44 score)
Chemotherapy-induced peripheral neurotoxicity as assessed by change in TNSn© scale | 5 YEARS
  difference between baseline and end of treatment of chemotherapy-induced peripheral neurotoxicity as assessed by change in TNSn© (changes from base line to end treatment of a 0-20 score)
Chemotherapy-induced peripheral neurotoxicity as assessed by change in PGIC scale | 5 YEARS
  difference between baseline and end of treatment of chemotherapy-induced peripheral neurotoxicity as assessed by change in PGIC (changes from base line to end treatment of a 0-10 score)
Chemotherapy-induced peripheral neurotoxicity as assessed by change in OXA-NQ scale | 5 YEARS
  difference between baseline and end of treatment of chemotherapy-induced peripheral neurotoxicity as assessed by change in OXA-NQ (changes from base line to end treatment of number of symptoms: this is a yes/no questionnaire for the presence of neuropathy symptoms)

SECONDARY OUTCOMES:
Chemotherapy-induced peripheral neurotoxicity as assessed by change in EORTC CIPN15 scale | 7 YEARS
  difference between baseline and end of treatment of chemotherapy-induced peripheral neurotoxicity as assessed by change in EORTC CIPN15 (changes of the global score of this questionnaire, 0-60)
Chemotherapy-induced peripheral neurotoxicity as assessed by change in TNSc© scale | 7 YEARS
  difference between baseline and end of treatment of chemotherapy-induced peripheral neurotoxicity as assessed by change in TNSc© (changes of the global score of this physician base scale ranging 0-48)
Chemotherapy-induced peripheral neurotoxicity as assessed by change in nerve conduction studies | 7 YEARS
  difference between baseline and end of treatment of chemotherapy-induced peripheral neurotoxicity as assessed by change in nerve conduction study of the radial (motor and sensory), ulnar (motor and sensory), sural, dorsal sural and common peroneal nerves. Amplitude (microV for sensory and mV for motor recordings) and velocity (m/sec) will be obtained. A decrease under the normative values at all time points respect to base line will be considered as sign of neuropathy.
Chemotherapy-induced peripheral neurotoxicity as assessed by change in Quantitative sensory testing (QST) | 7 YEARS
  difference between baseline and end of treatment of chemotherapy-induced peripheral neurotoxicity as assessed by change in QST: scores in seconds for time to pain onset and pain intensity (0=no pain; 10=worst pain
Chemotherapy-induced peripheral neurotoxicity as assessed by change in neurofilament light chain (NfL) levels | 7 YEARS
  difference between baseline and end of treatment of chemotherapy-induced peripheral neurotoxicity as assessed by change in Serum for biomarkers search: NfL dosage (pg/mL)
Chemotherapy-induced peripheral neurotoxicity as assessed by change in DN4 scale | 7 YEARS
  difference between baseline and end of treatment of chemotherapy-induced peripheral neurotoxicity as assessed by change in DN4 (this is a scale ranging 0-10)

CONTACTS AND LOCATIONS:
Overall Officials: GUIDO CAVALETTI, MD, Study Chair — University of Milano Bicocca; PAOLA ALBERTI, MD, Principal Investigator — University of Milano Bicocca
Locations (30):
- United States (8):
  - Birmingham School of Nursing, University of Alabama, Birmingham, Alabama
  - Northside Hospital, Atlanta, Georgia
  - JHU, Baltimore, Maryland
  - University of Michigan School of Nursing, Ann Arbor, Michigan
  - Columbia University Irving Medical Center, New York, New York
  - Cancer Center/Wexner Medical Center - Ohio State Medical Oncology Division, Columbus, Ohio
  - Dartmouth-Hitchcock Medical Center, Lebanon, Pennsylvania
  - University of Vermont Medical Center, Burlington, Vermont
- Brain and Mind Center, Sydney, Australia
- Dept. of Neurology, Medical University of Vienna, Vienna, Austria
- International Centre for Diarrhoeal Disease Research, Dhaka, Bangladesh
- Clínica AMO, Salvador, Brazil
- The Ottawa Hospital, Ottawa, Canada
- Aarhus University Hospital, Aarhus, Denmark
- France (2):
  - Hôpital Percy, Clamart
  - CHU Dupuytren, Limoges
- Center for Molecular Medicine, Cologne, Germany
- Greece (2):
  - University of Larissa, Larissa
  - "Saint Andrew's" State General Hospital, Pátrai
- Italy (6):
  - San Gerardo Hospital, Monza, Mb
  - Ospedale Valduce, Como
  - Ospedale Policlinico San Martino, Genova
  - A.O.U. Policlinico "G. Martino", Messina
  - Padova Hospital, Padua
  - Azienda Ospedaliera Universitaria, Verona
- Medical Oncoloy Unit - University of Nairobi, Nairobi, Kenya
- Centro Hospitalar Vila Nova de Gaia/Espinho, Vila Nova de Gaia, Portugal
- Dong-A University - Internal Medicine Dept., Busan, South Korea
- Hospital Universitari de Bellvitge-ICO L'Hospitalet, Barcelona, Spain
- University of Basel - Department of Sport, Exercise and Health, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No